CLINICAL TRIAL: NCT01069991
Title: Educating Adolescents To Preventively Manage Their Asthma
Brief Title: Asthma Self-Management For Adolescents
Acronym: ASMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York City Council Speaker's Fund (Unknown)
Responsible Party: Principal Investigator, David Evans PhD, Professor of Emeritus of Clinical Sociomedical Sciences (In Pediatrics) & Special Lecturer, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAB2642; R18HL67268 (Other Grant/Funding Number: New York City Council Speaker's Fund)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: Asthma; Adolescents; Patient Education; Schools
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient education group (Experimental): Patient education program delivered to high school students with persistent asthma.
  Interventions: Behavioral: Patient education group
- Wait list control group (Experimental): Control students received no intervention until the one year follow up period was completed.
  Interventions: Behavioral: Wait list control group

INTERVENTIONS:
Behavioral: Patient education group — Patient education delivered to high school students with persistent asthma in group and individual sessions. Academic detailing was also provided to the students' primary care providers.
  Arms: Patient education group
Behavioral: Wait list control group — No intervention was provided for this group until the one year study period was completed, and then the patient education intervention was provided.
  Arms: Wait list control group

SUMMARY:
The goal of this study is to help adolescents with asthma learn to control their illness and live without restrictions. We hypothesize that an intensive school-based asthma education program for students in 9th and 10th grade who have persistent asthma, together with asthma education for their primary care physicians, will improve the students' health status, quality of life, and ability to control their asthma through self-management.

DETAILED DESCRIPTION:
Five public high schools from areas in New York City with high asthma rates will be enrolled in the study. In each school, we will identify students with asthma using a brief, self-administered survey that asks questions about current symptoms of wheeze, persistent cough, chest tightness, night waking, and past diagnosis of asthma. Eligible students will have the program explained to them individually. Caregivers of students who express interest in the program will be contacted to obtain written, informed consent. An equal number of students in each school will be randomly assigned to the immediate intervention group and to a control group that will receive the program 12 months later. Students assigned to the immediate intervention group will take part in three group workshops to learn about the chronic nature of asthma, how to control asthma by monitoring symptoms and using medicines consistently, and how to take preventive management steps using environmental control strategies and a written treatment plan from their physician as a guide for adjusting their medicines. They will also receive individual coaching by a health educator to assess how the students are doing and feeling, help them interpret their symptoms and responses to medication, and encourage them to take the next steps to control asthma. Before the visit we will have asthma specialist physicians on our staff make a telephone call to the student's physician to alert them that the student will make a visit, that the student will bring symptoms diaries, and to encourage the physician to review the diaries, prescribe according to NHLBI guidelines, and provide a written treatment plan. The intervention for each student will last three months. During the follow up year, no educational contact will be made with control group students, families, or physicians. Following completion of the study 12 months later, these students will be offered the same intervention provided to the immediate intervention group.

ELIGIBILITY:
Inclusion Criteria:

* 9th or 10th grade high school student
* diagnosed moderate to severe persistent asthma
* used physician prescribed asthma medicine in past 12 months

Exclusion Criteria:

* comorbidity with other diseases that affect lung function
* enrollment in special education classes for learning disabilities

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 345 (Actual)
Dates: Start 2002-01; Primary Completion 2006-04 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Quality of life | One year

SECONDARY OUTCOMES:
Emergency department visits for asthma | One year

CONTACTS AND LOCATIONS:
Overall Officials: David Evans, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Bruzzese JM, Bonner S, Vincent EJ, Sheares BJ, Mellins RB, Levison MJ, Wiesemann S, Du Y, Zimmerman BJ, Evans D. Asthma education: the adolescent experience. Patient Educ Couns. 2004 Dec;55(3):396-406. doi: 10.1016/j.pec.2003.04.009. PMID 15582346